CLINICAL TRIAL: NCT02794857
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of NP001 in Subjects With Amyotrophic Lateral Sclerosis (ALS) and Evidence of Elevated Systemic Inflammation
Brief Title: Safety and Efficacy Study of NP001 in Patients With Amyotrophic Lateral Sclerosis (ALS) and Systemic Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuraltus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP001-10-003
Record Dates: First submitted 2016-05-24; First posted 2016-06-09 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neuromuscular Diseases; Inflammation; C-Reactive Protein
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neuromuscular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NP001 (Experimental): NP001 2 mg/kg by intravenous administration for 5 consecutive days in Month 1 and for 3 consecutive days in Months 2 through 6
  Interventions: Drug: NP001
- Placebo (Placebo Comparator): Normal saline by intravenous administration for 5 consecutive days in Month 1 and for 3 consecutive days in Months 2 through 6
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NP001
  Arms: NP001
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates NP001 in patients with amyotrophic lateral sclerosis (ALS) and evidence of systemic inflammation. Half of participants will receive NP001 and the other half will receive placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of NP001 in subjects with ALS and evidence of elevated systemic inflammation. Subjects will be allocated (1:1) to NP001 and placebo. Drug or placebo will be given intravenously.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of clinically possible, clinically probable (with or without laboratory support), or clinically definite ALS (using the revised El Escorial Criteria)
* Forced vital capacity greater than or equal to 65% of that predicted for age and height
* Onset of ALS-related weakness less than 3 years prior to first dose of study drug
* Plasma high sensitivity C-reactive protein (hs-CRP) concentration of greater than or equal to 0.113 mg/dL at pre-screening/screening
* Stable dose (greater than 30 days) of riluzole if undergoing treatment with this agent
* For females: Not be of childbearing potential or agree to use adequate birth control during the study

Key Exclusion Criteria:

* Life expectancy of less than 6 months
* Tracheotomy or be using ventilatory assistance, including Bi-level Positive Airway Pressure (BiPAP) or Continuous Positive Airway Pressure (CPAP)
* Active pulmonary disease
* Gastrostomy
* Stem cell therapy
* Immune modulator therapy or participation in studies of other agents within 12 weeks of pre-screening/screening
* Unstable medical condition other than ALS

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in score on ALS Functional Rating Scale-Revised (ALSFRS-R) questionnaire | Baseline and 6 months

SECONDARY OUTCOMES:
Change in pulmonary function as measured by slow vital capacity readings | Baseline and 6 months
Time to tracheotomy | Up to 6 months
Change in levels of blood inflammatory biomarkers | Baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gil Block, MD, PhD, Study Director — Neuraltus Pharmaceuticals, Inc.; Robert G. Miller, MD, Principal Investigator — California Pacific Medical Center; Jonathan Katz, MD, Principal Investigator — California Pacific Medical Center
Locations (22):
- United States (21):
  - St. Joseph's Hospital and Medical Center - Barrow Neurology Clinics, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Irvine, Department of Neurology, Orange, California
  - Forbes Norris MDA/ALS Research Center, CPMC, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Emory University, Department of Neurology, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Albert B. Chandler Medical Center, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Clinical & Translational Science Institute, University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Neurosciences Instutite-Neurology, Charlotte, North Carolina
  - Duke Neurological Disorders Clinic at Morreene Road, Durham, North Carolina
  - Cleveland Clinic Foundation-Cleveland Clinic Hospital, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Brain & Spine Institute, ALS Center, Portland, Oregon
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Texas Health Sciences Center San Antonio, San Antonio, Texas
- Montreal Neurological Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Forrest BD, Goyal NA, Fleming TR, Bracci PM, Brett NR, Khan Z, Robinson M, Azhir A, McGrath M. The Effectiveness of NP001 on the Long-Term Survival of Patients with Amyotrophic Lateral Sclerosis. Biomedicines. 2024 Oct 16;12(10):2367. doi: 10.3390/biomedicines12102367. PMID 39457678